CLINICAL TRIAL: NCT02568358
Title: DNA-based Testing in BAL of Lung Transplant Recipients With Suspected Non-viral Lower Respiratory Tract Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Thomas Fuehner, PD Dr. med. Thomas Fühner, Hannover Medical School
Other Study IDs: LuTx_Mibi-DNA-1
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Lower Respiratory Tract and Lung Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchoalveolar lavage
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Experimental Intervention: DNA-based testing of BAL fluid — DNA based testing needs 4.5 hours lab time in addition to standard testing

SUMMARY:
Lung transplantation (LTx) , DNA-based testing.

Performance of DNA-based testing of bacterial and fungal pathogens in comparison to standard testing.

Experimental intervention: DNA-based testing of BAL fluid.

DETAILED DESCRIPTION:
Cohen's kappa of any pathogen isolation by DNA-based testing vs. standard cultures in comparison to the final diagnosis of non-viral lower respiratory tract infection.

ELIGIBILITY:
Inclusion Criteria:

* patients after lung transplantation (single, double or combined)
* suspicion of non-viral lower respiratory tract infection as defined by at least 2 out of
* new onset of malaise
* new or progressive pulmonary infiltrate
* hypoxemia (SpO2/SaO2 <92% or need for oxygen)
* temperature of 38 o C or above within 7 days
* purulent (yellow or greenish) sputum
* CRP of 30 mg/l or above
* PCT of 0,5 µg/l or above

Exclusion Criteria:

* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant recipients with suspected non-viral lower respiratory tract infection
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Cohen's kappa of any pathogen isolation by DNA-based testing vs. standard cultures in comparison to the final diagnosis of non-viral lower respiratory tract infection | 6 month
  Cohen's kappa measures the agreement between methods and the final clinical diagnosis. Both methods (DNA-based testing and standard cultures) will result in isolation of a non-viral pathogen or no isolation of a pathogen. A final clinical diagnosis will classify patients clinically in two categories as non-viral lower respiratory tract infection or no non-viral lower respiratory tract infection usually made 48-72 hours made after sampling. Cohen's kappa will be compared between the two methods.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gottlieb, Prof. Dr., Principal Investigator — Hannover Medical School